CLINICAL TRIAL: NCT05180253
Title: Healthy Control Esophageal and Gastric Registry and Biorepository
Brief Title: Esophageal and Gastric Registry and Biorepository
Status: Recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Benjamin D Rogers, Assistant Professor, M.D., University of Louisville
Other Study IDs: 20.0990
Record Dates: First submitted 2021-10-28; First posted 2022-01-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Gastro Esophageal Reflux
Keywords: Mucosal Integrity; Functional Luminal Imaging Probe
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Up to 10 research biopsies will be taken from the sides of your esophagus. An additional 2 research biopsies will be taken from the stomach. Additional esophageal biopsies may be taken at the discretion of the gastroenterologist performing the endoscopy if clinically indicated to be analyzed by the hospital's pathology department.
  Each biopsy taken for research purposes will be processed and stored by a code that will not contain any personal information.
  Samples of tissue from the esophageal biopsy will also be frozen and stored for future unspecified research, including comparing them to other disease populations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Subjects
  Interventions: Diagnostic Test: Esophageal studies

INTERVENTIONS:
Diagnostic Test: Esophageal studies — Healthy subjects will undergo esophageal and blood testing.

SUMMARY:
The evaluation of the foregut, the esophagus and stomach, has come a long way over the past two decades, and continues to experience exciting discoveries in the clinical evaluation of foregut physiology. Assessing esophageal peristalsis has relied for the past several decades on High Resolution Manometry (HRM), however it has recently become known that even though HRM is an extremely effective tool, that there are certain subsets of patients in which additional information is required. Additionally, the assessment of esophageal reflux disease has relied on pH impedance for the last two decades. However, this procedure requires a catheter to be passed through a nostril and remain in place for at least 24 hours. Novel techniques, already FDA approved, including EndoFLIP for esophageal peristalsis and mucosal integrity (MI) for reflux disease, have emerged as time-of-endoscopy assessments. Both involve the placement of a balloon through the scope at time of upper endoscopy (standard first line assessment for both dysphagia and reflux symptoms) and are quick and pose little-to-no additional risk or discomfort for patients. However, data regarding normal esophageal parameters are poorly defined for both EndoFLIP and MI. Additionally, EndoFLIP has increasingly been used to assess the pylorus, and scarce data exists there regarding how a tool originally envisioned for esophageal assessment can be used more distally in the GI tract.

We will recruit healthy, asymptomatic volunteers to undergo testing with MI and FLIP (esophageal and pyloric). The data obtained will help establish the benchmark from which assessments can be made in patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* No prior surgical history
* Asymptomatic according to gastroesophageal and gastric questionnaires
* Not currently taking any medications that affect acid secretion or gut motility
* No history of malignancy
* No mental health issues precluding informed consent
* No smoking history
* No excessive or daily alcohol use
* BMI < 30
* No known hiatus hernia
* No known medical illness (autoimmune, neurological) that could be associated with altered esophageal or gastric function
* Not allergic to fentanyl or versed
* No history of eating disorder
* No history of autoimmune disorders

Exclusion Criteria:

* Minors
* Surgeries involving the GI tract
* Medication use affecting acid secretion or gut motility
* Personal history of malignancy
* Mental health issues precluding informed consent
* Symptoms on standard clinical questionnaires
* Pregnant - the effect that pregnancy has on esophageal and gastric motility is not well defined, but we will need to eliminate this as a confounding factor
* Nursing women - although the investigations are FDA approved and part of standard clinic practices, they are time consuming and involve medication administration that might affect the ability of a mother to nurse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18-85 years of age, free of esophageal symptoms, never diagnosed with esophageal disorders, never diagnosed with an autoimmune disease, able to provide informed consent, and willing and able to undergo esophageal physiologic studies and biopsies.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Normative mucosal integrity values | 1 year
  We will establish the range of MI values in healthy, asymptomatic individuals.
Normative pyloric FLIP values | 1 year
  We will further establish the range of FLIP values that can be seen in healthy, asymptomatic individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Norton Healthcare, Louisville, Kentucky, United States